CLINICAL TRIAL: NCT04281745
Title: A Single-arm Trial, Open-label, Repeated, Long-term, Multi-center, Phase IV Clinical Trial to Evaluate the Long-term Efficacy and Safety of Repeat Treatment of Glabellar Lines With CORETOX®
Brief Title: Long-term Open-label Treatment of Moderate to Severe Glabellar Lines With CORETOX®
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT03-KR19GBL404
Record Dates: First submitted 2020-02-17; First posted 2020-02-24 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coretox® (Experimental): Botulinum toxin type A to be intramuscularly injected at 4 sites of corrugator muscle and at 1 site of procerus muscle with 0.1 mL (4U) at each site, for a total of 0.5 mL (20U). The administration of the investigational product was performed once at the start of each cycle
  Interventions: Biological: CORETOX Inj

INTERVENTIONS:
Biological: CORETOX Inj — Clostridium botulinum type A (Hall group); a lyophilized white power for injection with a colorless transparent vial. colorless transparent solution when dissolved with saline.
  Other Names: Botulinum toxin type A

SUMMARY:
This study evaluates the long-term safety and efficacy of CORETOX in the treatment of moderate to severe glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 20 and 65
* Patients attaining ≥grade 2 (moderate) in the investigator's rating of the severity of glabella lines at maximum frown
* Patients who can comply with the study procedures and visit schedule
* Patients who voluntarily sign the informed consent

Exclusion Criteria:

* Patients with medical conditions who may be at greater risk due to the administration of the investigational drugs (e.g.. diseases that may affect the neuromuscular action including Myasthenia Gravis, Lambert-Eaton Syndrome, Amyotrophic Lateral Sclerosis and motor neuropathy)
* Patients with the history of facial nerve paralysis or the symptoms of eyelid ptosis
* Patients who have received other procedures which may affect glabellar and forehead lines within 6 months
* Patients who have received other procedures which may affect glabellar and forehead lines within 6 months
* Patients who were injected with botulinum toxin within the past 3 months
* Patients with allergy or hypersensitivity to the investigational drugs or their components
* Patients who have bleeding tendency or taking anti-coagulant
* Female subjects who are pregnant or lactating. Female subjects of childbearing age who have a plan to get pregnant during the study period, or do not use available contraceptive methods (Women of childbearing age should have negative urine pregnancy test results at baseline visit (0 week) prior to the first injection.)
* Patients with skin disorders or infection at the injection site
* Patients who are participating in other clinical trials or have participated in other clinical trials 30 days before screening
* Patients who are unable to communicate or follow the instructions
* Patients who are not eligible for this study based on the judgment of an investigator

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2022-03-16 (Estimated)

PRIMARY OUTCOMES:
Investigator-rated improvement rate of glabellar lines at maximum frown at Week 4 of each treatment cycle | At Week 4 of each cycle (each cycle lasts until re-treatment, where re-treatment is possible after 90 Days from the last treatment).
  Improvement rate: improvement of Facial Wrinkle Scale score from 3 (moderate) or 4 (severe) to 0 (none) or 1 (mild)
Subject-rated improvement rate of glabellar lines at maximum frown | Every 4 weeks in each treatment cycle (each cycle lasts until re-treatment, where re-treatment is possible after 90 Days from the last treatment).
Subject-rated satisfaction at each cycle after treatment | Every 4 weeks in each treatment cycle (each cycle lasts until re-treatment, where re-treatment is possible after 90 Days from the last treatment).
Treatment on-set date | From baseline to Day 7 of each cycle (each cycle lasts until re-treatment, where re-treatment is possible after 90 Days from the last treatment).
Treatment duration | From on-set date to next treatment (each cycle lasts until re-treatment, where re-treatment is possible after 90 Days from the last treatment).
Number of participants who experienced an adverse event | Baseline to Day 720
Number of participants with binding and neutralizing antibodies | Screening and Day 720

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea